CLINICAL TRIAL: NCT00408629
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Study of the Human Anti-TNF Monoclonal Antibody Adalimumab for the Induction and Maintenance of Clinical Remission in Subjects With Moderately to Severely Active Ulcerative Colitis
Brief Title: Efficacy and Safety of Adalimumab in Subjects With Moderately to Severely Active Ulcerative Colitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Roopal B Thakker, M.D./Project Director, Abbott
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M06-827; 2006-002782-40 (EudraCT Number)
Record Dates: First submitted 2006-12-05; First posted 2006-12-07 (Estimated); Results first posted 2011-03-31 (Estimated); Last update posted 2011-05-03 (Estimated); Status verified 2011-04

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative Colitis; Adalimumab; TNF Antagonist; Mayo Score
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- adalimumab group (Experimental)
  Interventions: Biological: adalimumab
- placebo group (Experimental)
  Interventions: Biological: placebo

INTERVENTIONS:
Biological: adalimumab — Prefilled syringe, 40 mg, 160 mg at Week 0, 80 mg at Week 2, and 40 mg every other week between Weeks 4 and 50.
  Other Names: ABT-D2E7; Humira
  Arms: adalimumab group
Biological: placebo — Matching Placebo for prefilled syringe, 40 mg,
  Arms: placebo group

SUMMARY:
This was a Phase 3, multicenter, randomized, double-blind, placebo-controlled trial designed to evaluate the efficacy and safety of the human anti-tumor necrosis factor (TNF) monoclonal antibody adalimumab (ADA) in patients with moderately to severely active ulcerative colitis (UC).

DETAILED DESCRIPTION:
This was a Phase 3, multicenter, randomized, double-blind, placebo-controlled trial designed to evaluate the efficacy and safety of adalimumab (ADA) in patients with moderately to severely active ulcerative colitis (UC).

The duration of the study was up to 65 weeks, including a Screening Period of up to 3 weeks, a double-blind (DB) placebo-controlled treatment period of up to 52 weeks, and a 70 day follow-up phone call for participants who prematurely discontinued or who did not enroll in the extension study NCT# 00573794 (M10-223).

Adult participants with moderate to severe UC (Mayo score of 6 to 12 points with endoscopy subscore of 2 to 3 points), confirmed by colonoscopy with biopsy or flexible sigmoidoscopy with biopsy, were to be enrolled at approximately 120 sites worldwide. Planned enrollment was 500 participants.

Participants were to be stratified by prior exposure to infliximab and/or other anti-TNF agents, and randomized in a 1:1 ratio to receive ADA or placebo by subcutaneous injection. Participants assigned to the ADA treatment arm were to receive an induction dose of 160 mg at Week 0 and 80 mg at Week 2, and 40 mg every other week (eow) starting at Week 4. Participants assigned to the placebo treatment arm were to receive matching placebo during the same period of time. At or after Week 10, participants who met the criteria for inadequate response could be switched to open-label (OL) ADA 40 mg eow beginning at Week 12. Inadequate response was defined as:

* Partial Mayo score greater than or equal to Baseline score on 2 consecutive visits at least 14 days apart (for participants with a partial Mayo score of 4 to 7 at Baseline).
* Partial Mayo score greater than or equal to 7 on 2 consecutive visits at least 14 days apart (for participants with a partial Mayo score of 8 or 9 at Baseline).

Participants who demonstrated inadequate response at 2 consecutive visits at least 14 days apart while on OL administration ADA 40 mg eow were permitted to dose escalate to ADA 40 mg weekly (ew). Participants with persistent inadequate response while on ADA 40 mg ew may have been discontinued from the study at the Investigator's discretion. Upon completion of the study, participants had the option to enroll into the OL extension Study M10-223 in which they could receive ADA treatment.

Efficacy and safety measurements were performed throughout the study. A follow-up phone call was made 70 days after the last dose of study drug to obtain information on any ongoing or new adverse events (AEs) for all participants who terminated early or who did not enroll in the OL extension study.

ELIGIBILITY:
Inclusion Criteria:

1. Participants >=18 years of age and in good health (Investigator discretion) with a recent stable medical history
2. Diagnosis of UC for greater than 90 days prior to Baseline
3. Diagnosis of active UC confirmed by colonoscopy with biopsy or flexible sigmoidoscopy with biopsy during the Screening Period, with exclusion of infection
4. Active UC with a Mayo score of 6 to 12 points and endoscopy subscore of 2 to 3 points, despite concurrent treatment with at least 1 of the following (oral corticosteroids or immunosuppressants or both as defined below):

   * Stable oral corticosteroid dose (prednisone >= 20 mg/day or equivalent) for at least 14 days prior to Baseline or maintenance, corticosteroid dose (prednisone < 20 mg/day or equivalent) for at least 40 days prior to Baseline

   and/or
   * At least a 90 day course of azathioprine (AZA) or 6-mercaptopurine (6-MP) prior to Baseline, with a dose of AZA >= 1.5 mg/kg/day or 6-MP >= 1 mg/kg/day (rounded to the nearest available tablet formulation), or a dose that is the highest tolerated by the participant (e.g., due to leukopenia, elevated liver enzymes, nausea) during that time. Participant must be on a stable dose for at least 28 days prior to Baseline.

   Concurrent therapy was not required for participants who were previously treated with corticosteroids or immunosuppressants (AZA or 6-MP) during the past 5 years and in the judgment of the Investigator have failed to respond to, or could not tolerate, their treatment.
5. Participants may have been included if they had previously used an anti-tumor necrosis factor (TNF) agent (except ADA) and discontinued its use due to a loss of response or intolerance to the agent.
6. Had to be able to self-administer or had caregiver who could reliably administer subcutaneous (SC) injections.
7. Had to be able and willing to give written informed consent and to comply with the requirements of the study protocol.
8. Female had to be either not of childbearing potential, defined as postmenopausal for at least 1 year or surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy), or of childbearing potential and practicing an approved method of birth control throughout the study and for 150 days after the last dose of study drug. Examples of approved methods of birth control included the following:

   * Condoms, sponge, foams, jellies, diaphragm, or intrauterine device
   * Oral, parenteral, intravaginal contraceptives for 90 days prior to study drug administration
   * A vasectomized partner The results of the serum pregnancy test performed at the Screening Visit and urine pregnancy test performed at the Baseline Visit must have been negative.
9. Judged to be in generally good health as determined by the Investigator

Exclusion Criteria:

1. History of subtotal colectomy with ileorectostomy or colectomy with ileoanal pouch, Koch pouch, or ileostomy for UC, or planned bowel surgery.
2. Received previous treatment with ADA or previous participation in an ADA clinical study.
3. Received cyclosporine, tacrolimus, or mycophenolate mofetil within 30 days of Baseline.
4. Received intravenous (IV) corticosteroids within 14 days of Screening or during the Screening Period.
5. Received therapeutic enema or suppository, other than required for endoscopy, within 14 days of the Screening endoscopy and during the remainder of the Screening Period.
6. Current diagnosis of fulminant colitis and/or toxic megacolon.
7. Disease limited to the rectum (ulcerative proctitis).
8. Current diagnosis of indeterminate colitis.
9. Current diagnosis and/or history of Crohns disease (CD).
10. Currently receiving total parenteral nutrition.
11. Used aminosalicylates for < 90 days before Baseline or not on a stable dose for at least 28 days before Baseline or discontinued use within 28 days of Baseline.
12. Positive Clostridium difficile stool assay.
13. Previously used infliximab or any anti-TNF agent within 56 days of Baseline.
14. Previously used infliximab or any anti-TNF agent without clinical response at any time ("primary non-responder") unless subject experienced a treatment-limiting reaction.
15. Infections requiring treatment with IV antibiotics, antivirals, or antifungals within 30 days of Baseline or oral antibiotics, antivirals, or antifungals within 14 days of Baseline.
16. History of malignancy other than a successfully treated non-metastatic cutaneous squamous cell or basal cell carcinoma and/or localized carcinoma in situ of the cervix. If the Screening colonoscopy/flexible sigmoidoscopy showed evidence of dysplasia or a malignancy, subject was not to be enrolled in the study.
17. History of listeria, histoplasmosis, chronic or active hepatitis B infection, human immunodeficiency virus (HIV), immunodeficiency syndrome, central nervous system demyelinating disease, or untreated tuberculosis (TB).
18. Female subject who was pregnant or breast-feeding or considering becoming pregnant during the study (there should be at least 150 days between the last dose of study drug and either conception or initiation of breast-feeding in women of childbearing potential).
19. Poorly controlled medical condition(s), such as uncontrolled diabetes, unstable ischemic heart disease, moderate to severe congestive heart failure (CHF), recent cerebrovascular accident, and any other condition, which in the opinion of the investigator, put the subject at risk by participation in the protocol.
20. Received any investigational agent within 30 days or 5 half lives prior to Baseline (whichever was longer).
21. History of clinically significant drug or alcohol abuse during the past year.
22. Known hypersensitivity to the excipients of ADA as stated in the label.
23. Any prior exposure to Tysabri® (natalizumab), or Orencia® (abatacept) or any other biological therapy [other than Kineret® (anakinra) and anti-TNF agents].
24. Currently taking both budesonide and prednisone (or equivalent) simultaneously.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 518 (Actual)
Dates: Start 2006-11; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roopal B Thakkar, M.D., Study Director — Abbott
Locations (108):
- United States (36):
  - Site Ref # / Investigator 5394, Anaheim, California
  - Site Ref # / Investigator 3753, Wheat Ridge, Colorado
  - Site Ref # / Investigator 3754, Hamden, Connecticut
  - Site Ref # / Investigator 12903, Gainesville, Florida
  - Site Ref # / Investigator 3747, Hollywood, Florida
  - Site Ref # / Investigator 5106, Jacksonville, Florida
  - Site Ref # / Investigator 11601, Naples, Florida
  - Site Ref # / Investigator 6846, Sarasota, Florida
  - Site Ref # / Investigator 3742, Winter Park, Florida
  - Site Ref # / Investigator 3760, Zephyrhills, Florida
  - Site Ref # / Investigator 3739, Atlanta, Georgia
  - Site Ref # / Investigator 7658, Macon, Georgia
  - Site Ref # / Investigator 5397, Moline, Illinois
  - Site Ref # / Investigator 7453, Topeka, Kansas
  - Site Ref # / Investigator 3759, Annapolis, Maryland
  - Site Ref # / Investigator 3762, Annapolis, Maryland
  - Site Ref # / Investigator 3738, Lutherville, Maryland
  - Site Ref # / Investigator 7472, Troy, Michigan
  - Site Ref # / Investigator 3744, Rochester, Minnesota
  - Site Ref # / Investigator 6088, St Louis, Missouri
  - Site Ref # / Investigator 3756, Great Neck, New York
  - Site Ref # / Investigator 3752, Charlotte, North Carolina
  - Site Ref # / Investigator 3758, Jacksonville, North Carolina
  - Site Ref # / Investigator 3745, Cincinnati, Ohio
  - Site Ref # / Investigator 7709, Oklahoma City, Oklahoma
  - Site Ref # / Investigator 3740, Tulsa, Oklahoma
  - Site Ref # / Investigator 3765, Sayre, Pennsylvania
  - Site Ref # / Investigator 3741, Columbia, South Carolina
  - Site Ref # / Investigator 3737, Germantown, Tennessee
  - Site Ref # / Investigator 6077, Nashville, Tennessee
  - Site Ref # / Investigator 5107, Nashville, Tennessee
  - Site Ref # / Investigator 3743, Nashville, Tennessee
  - Site Ref # / Investigator 5398, Ogden, Utah
  - Site Ref # / Investigator 8064, Spokane, Washington
  - Site Ref # / Investigator 3750, Spokane, Washington
  - Site Ref # / Investigator 3761, West Bend, Wisconsin
- Site Ref # / Investigator 6853, Buenos Aires, Argentina
- Australia (7):
  - Site Ref # / Investigator 13722, Garran, Australian Capital Territory
  - Site Ref # / Investigator 16141, Bankstown, New South Wales
  - Site Ref # / Investigator 13723, Herston, Queensland
  - Site Ref # / Investigator 10706, Bedford Park, South Australia
  - Site Ref # / Investigator 14882, Box Hill, Victoria
  - Site Ref # / Investigator 9002, Malvern, Victoria
  - Site Ref # / Investigator 10704, Fremantle, Western Australia
- Site Ref # / Investigator 9802, Vienna, Austria
- Belgium (5):
  - Site Ref # / Investigator 5256, Bonheiden
  - Site Ref # / Investigator 5253, Brussels
  - Site Ref # / Investigator 6225, Brussels
  - Site Ref # / Investigator 6079, Ghent
  - Site Ref # / Investigator 6078, Leuven
- Canada (9):
  - Site Ref # / Investigator 10423, Kelowna, British Columbia
  - Site Ref # / Investigator 3766, Victoria, British Columbia
  - Site Ref # / Investigator 13556, Greater Sudbury, Ontario
  - Site Ref # / Investigator 3769, Hamilton, Ontario
  - Site Ref # / Investigator 3736, Toronto, Ontario
  - Site Ref # / Investigator 3771, Montreal, Quebec
  - Site Ref # / Investigator 3764, Montreal, Quebec
  - Site Ref # / Investigator 3768, Montreal, Quebec
  - Site Ref # / Investigator 3770, Québec, Quebec
- Czechia (5):
  - Site Ref # / Investigator 7021, České Budějovice
  - Site Ref # / Investigator 6307, Hradec Kravlove 12
  - Site Ref # / Investigator 6606, Olomouc
  - Site Ref # / Investigator 7481, Prague
  - Site Ref # / Investigator 7479, Prague
- Denmark (2):
  - Site Ref # / Investigator 6483, Hvidovre
  - Site Ref # / Investigator 7477, Odense C
- France (4):
  - Site Ref # / Investigator 6231, Clichy
  - Site Ref # / Investigator 7476, Lille
  - Site Ref # / Investigator 7475, Pessac
  - Site Ref # / Investigator 7474, Toulouse
- Germany (8):
  - Site Ref # / Investigator 15321, Hamburg
  - Site Ref # / Investigator 9069, Hamburg
  - Site Ref # / Investigator 14642, Magdeburg
  - Site Ref # / Investigator 9067, Minden
  - Site Ref # / Investigator 14661, Munich
  - Site Ref # / Investigator 9801, Munich
  - Site Ref # / Investigator 14761, Münster
  - Site Ref # / Investigator 5247, Regensburg
- Hungary (6):
  - Site Ref # / Investigator 7485, Budapest
  - Site Ref # / Investigator 5025, Budapest
  - Site Ref # / Investigator 10625, Debrecen
  - Site Ref # / Investigator 14104, Gyula
  - Site Ref # / Investigator 4987, Miskoic
  - Site Ref # / Investigator 5036, Miskolc
- Israel (3):
  - Site Ref # / Investigator 12744, Kfar Saba
  - Site Ref # / Investigator 10623, Petah Tikva
  - Site Ref # / Investigator 15361, Tel Aviv
- New Zealand (4):
  - Site Ref # / Investigator 13301, Auckland
  - Site Ref # / Investigator 13181, Auckland
  - Site Ref # / Investigator 13148, Christchurch
  - Site Ref # / Investigator 13482, Hamilton
- Norway (5):
  - Site Ref # / Investigator 9561, Gjøvik
  - Site Ref # / Investigator 5197, Oslo
  - Site Ref # / Investigator 6297, Oslo
  - Site Ref # / Investigator 5194, Tromsø
  - Site Ref # / Investigator 5193, Trondheim
- Poland (4):
  - Site Ref # / Investigator 5242, Lodz
  - Site Ref # / Investigator 5266, Warsaw
  - Site Ref # / Investigator 5265, Warsaw
  - Site Ref # / Investigator 15263, Wroclaw
- Portugal (3):
  - Site Ref # / Investigator 5264, Faro
  - Site Ref # / Investigator 7473, Lisbon
  - Site Ref # / Investigator 5263, Lisbon
- Spain (2):
  - Site Ref # / Investigator 5211, Barcelona
  - Site Ref # / Investigator 5212, Madrid
- Switzerland (3):
  - Site Ref # / Investigator 10221, Basel
  - Site Ref # / Investigator 10222, Bern
  - Site Ref # / Investigator 9162, Zurich

REFERENCES:
- [Derived] Ryan C, Sobell JM, Leonardi CL, Lynde CW, Karunaratne M, Valdecantos WC, Hendrickson BA. Safety of Adalimumab Dosed Every Week and Every Other Week: Focus on Patients with Hidradenitis Suppurativa or Psoriasis. Am J Clin Dermatol. 2018 Jun;19(3):437-447. doi: 10.1007/s40257-017-0341-6. PMID 29380251
- [Derived] Wolf D, D'Haens G, Sandborn WJ, Colombel JF, Van Assche G, Robinson AM, Lazar A, Zhou Q, Petersson J, Thakkar RB. Escalation to weekly dosing recaptures response in adalimumab-treated patients with moderately to severely active ulcerative colitis. Aliment Pharmacol Ther. 2014 Sep;40(5):486-97. doi: 10.1111/apt.12863. Epub 2014 Jul 15. PMID 25041859
- [Derived] Feagan BG, Sandborn WJ, Lazar A, Thakkar RB, Huang B, Reilly N, Chen N, Yang M, Skup M, Mulani P, Chao J. Adalimumab therapy is associated with reduced risk of hospitalization in patients with ulcerative colitis. Gastroenterology. 2014 Jan;146(1):110-118.e3. doi: 10.1053/j.gastro.2013.09.032. Epub 2013 Sep 22. PMID 24067881
- [Derived] Sandborn WJ, Colombel JF, D'Haens G, Van Assche G, Wolf D, Kron M, Lazar A, Robinson AM, Yang M, Chao JD, Thakkar R. One-year maintenance outcomes among patients with moderately-to-severely active ulcerative colitis who responded to induction therapy with adalimumab: subgroup analyses from ULTRA 2. Aliment Pharmacol Ther. 2013 Jan;37(2):204-13. doi: 10.1111/apt.12145. Epub 2012 Nov 23. PMID 23173821

RESULTS

PARTICIPANT FLOW:
Groups:
- Adalimumab 160/80/40: During the Double-Blind (DB) period, the Adalimumab (ADA) treatment group received a dose of 160 mg at Week 0, 80 mg at Week 2, and 40 mg every other week (eow) starting at Week 4 (160/80/40 mg).
- Placebo: The placebo treatment group received placebo throughout the Double-Blind (DB) period.
Period: Overall Study
Arm/Group | Adalimumab 160/80/40 | Placebo
Started | 258 (10 ADA recipients from 3 noncompliant clinical sites in Safety, but not in Efficacy analyses (248).) | 260 (14 PLB recipients from 3 noncompliant clinical sites in Safety, but not in Efficacy analyses (246).)
Completed | 161 (1 ADA recipient did not receive study drug and discontinued due to other reasons.) | 135
Not Completed | 97 | 125
Not completed — Adverse Event | 13 | 27
Not completed — Withdrawal by Subject | 8 | 4
Not completed — Lost to Follow-up | 1 | 1
Not completed — Lack of Efficacy | 63 | 73
Not completed — Protocol Violation | 1 | 5
Not completed — Miscellaneous | 11 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adalimumab 160/80/40 | Placebo | Total
Number analyzed (Participants) | 248 | 246 | 494
Age Continuous [Mean (Standard Deviation); unit: Years] — The ITT analysis set, defined as all participants who were randomized in the study excluding participants from 3 non-compliant sites, was used to determine all Baseline measures (continuous age, customized age, gender, and region of enrollment).
  Years | 39.6 (12.47) | 41.3 (13.22) | 40.4 (12.86)
Age, Customized [Number; unit: Participants]
  < 40 years | 136 | 118 | 254
  40 to 64 years | 105 | 116 | 221
  >=65 years | 7 | 12 | 19
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 106 | 94 | 200
  Male | 142 | 152 | 294
Region of Enrollment [Number; unit: Participants]
  Portugal | 2 | 1 | 3
  United States | 78 | 82 | 160
  Spain | 4 | 7 | 11
  Austria | 0 | 4 | 4
  Israel | 5 | 0 | 5
  France | 18 | 14 | 32
  Czech Republic | 18 | 25 | 43
  Hungary | 13 | 13 | 26
  Canada | 18 | 19 | 37
  Poland | 14 | 15 | 29
  Belgium | 26 | 18 | 44
  Australia | 11 | 9 | 20
  Denmark | 2 | 3 | 5
  Norway | 5 | 1 | 6
  Germany | 19 | 22 | 41
  New Zealand | 4 | 4 | 8
  Switzerland | 11 | 9 | 20

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Who Achieved Clinical Remission Per Mayo Score at Week 8
Description: Clinical remission per Mayo score is defined as a total Mayo score of at least 2 and no individual subscore greater than 1. The Mayo Score is a discrete ordinal scale ranging from 0 (normal or inactive disease) to 12 (severe disease) and is a composite of 4 subscores:
  Stool Frequency Subscore (SFS), Rectal Bleeding Subscore (RBS), Endoscopy Subscore, and Physician's Global Assessment Subscore (PGA), each of which ranges from 0 (normal) to 3 (severe disease).
Time Frame: Week 8
Population: Intent-to-treat (ITT) analysis set using the non-responder imputation (NRI) method in which all missing remission values and values after switch to open-label (OL) treatment were considered to be non-remission.
Measure: Number; unit: Percentage of Participants
Arm/Group | Adalimumab 160/80/40 | Placebo
Number analyzed (Participants) | 248 | 246
Percentage of Participants | 16.5 | 9.3
Statistical Analysis 1: Comparison: Adalimumab 160/80/40 vs Placebo; Assuming that 5% of the subjects in the placebo group achieve clinical remission at Week 52 or Week 8, a sample size of 250 in each treatment group will be adequate to detect a difference of at least 7 percentage points from the adalimumab group using Chi squared test with 80% power at a 0.05 two-sided significance level; Test type: Superiority or Other; p = 0.019, Cochran-Mantel-Haenszel — Testing for ranked co-primary endpoints occurred in hierarchical order to control for multiple testing. Week 8 remission rate was tested first. If a significant difference in group rates was found at alpha=0.05, Week 52 rate was tested at alpha=0.05; Stratification levels for Cochran-Mantel-Haenszel = prior anti-TNF versus anti-TNF-naive

2. Primary Outcome: Proportion of Participants Who Achieved Clinical Remission Per Mayo Score at Week 52
Description: Clinical remission per Mayo score is defined as a total Mayo score of at least 2 and no individual subscore greater than 1. The Mayo Score is a discrete ordinal scale ranging from 0 (normal or inactive disease) to 12 (severe disease) and is a composite of 4 subscores:
  SFS, RBS, Endoscopy Subscore, and PGA, each of which ranges from 0 (normal) to 3 (severe disease).
Time Frame: Week 52
Population: Intent-to-treat analysis set using the non-responder imputation (NRI) method in which all missing remission values and values after switch to OL treatment were considered to be non-remission.
Measure: Number; unit: Percentage of Participants
Arm/Group | Adalimumab 160/80/40 | Placebo
Number analyzed (Participants) | 248 | 246
Percentage of Participants | 17.3 | 8.5
Statistical Analysis 1: Comparison: Adalimumab 160/80/40 vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.004, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Stratification levels for Cochran-Mantel-Haenszel = prior anti-TNF versus anti-TNF-naive

3. Secondary Outcome: Proportion of Participants Who Achieved Sustained Clinical Remission Per Mayo Score at Both Week 8 and Week 52
Description: as for outcome 2
Time Frame: Week 8, Week 52
Population: Intent-to-treat analysis set using the non-responder imputation (NRI) method in which all missing remission values and values after switch to open-label treatment were considered to be non-remission.
Measure: Number; unit: Percentage of Participants
Arm/Group | Adalimumab 160/80/40 | Placebo
Number analyzed (Participants) | 248 | 246
Percentage of Participants | 8.5 | 4.1
Statistical Analysis 1: Comparison: Adalimumab 160/80/40 vs Placebo; The Cochran-Mantel-Haenszel test was used to test the null hypothesis of no difference between adalimumab and placebo. Treatment differences were deemed statistically significant at a significance level of 0.05; Test type: Superiority or Other; p = 0.047, Cochran-Mantel-Haenszel — Testing of ranked secondary measures was only started if significant group differences existed for both co-primary measures. Significant results for higher-ranked measure was needed to test next lower-ranked measure to control for multiple testing; Stratification levels for Cochran-Mantel-Haenszel = prior anti-TNF versus anti-TNF-naive

4. Secondary Outcome: Proportion of Participants Who Achieved Clinical Response Per Mayo Score at Week 8
Description: Clinical response per Mayo score is defined as a decrease in Mayo score of at least 3 points and at least 30% from Baseline, plus either a decrease in rectal bleeding subscore (RBS) of at least 1 point from Baseline or an absolute RBS of 0 or 1. The Mayo Score is a discrete ordinal scale ranging from 0 (normal or inactive disease) to 12 (severe disease) and is a composite of 4 subscores:
  SFS, RBS, Endoscopy Subscore, and PGA, each of which ranges from 0 (normal) to 3 (severe disease).
Time Frame: Week 8
Population: as for outcome 3
Measure: Number; unit: Percentage of Participants
Arm/Group | Adalimumab 160/80/40 | Placebo
Number analyzed (Participants) | 248 | 246
Percentage of Participants | 50.4 | 34.6
Statistical Analysis 1: Comparison: Adalimumab 160/80/40 vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; Stratification levels for Cochran-Mantel-Haenszel = prior anti-TNF versus anti-TNF-naive

5. Secondary Outcome: Proportion of Participants Who Achieved Clinical Response Per Mayo Score at Week 52
Description: Clinical response per Mayo score is defined as a decrease in Mayo score of at least 3 points and at least 30% from Baseline, plus either a decrease in RBS of at least 1 point from Baseline or an absolute RBS of 0 or 1. The Mayo Score is a discrete ordinal scale ranging from 0 (normal or inactive disease) to 12 (severe disease) and is a composite of 4 subscores:
  SFS, RBS, Endoscopy Subscore, and PGA, each of which ranges from 0 (normal) to 3 (severe disease).
Time Frame: Week 52
Population: as for outcome 3
Measure: Number; unit: Percentage of Participants
Arm/Group | Adalimumab 160/80/40 | Placebo
Number analyzed (Participants) | 248 | 246
Percentage of Participants | 30.2 | 18.3
Statistical Analysis 1: Comparison: Adalimumab 160/80/40 vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.002, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; Stratification levels for Cochran-Mantel-Haenszel = prior anti-TNF versus anti-TNF-naive

6. Secondary Outcome: Proportion of Participants Who Achieved Sustained Clinical Response Per Mayo Score at Both Week 8 and Week 52
Description: as for outcome 5
Time Frame: Week 8, Week 52
Population: as for outcome 3
Measure: Number; unit: Percentage of Participants
Arm/Group | Adalimumab 160/80/40 | Placebo
Number analyzed (Participants) | 248 | 246
Percentage of Participants | 23.8 | 12.2
Statistical Analysis 1: Comparison: Adalimumab 160/80/40 vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; Stratification levels for Cochran-Mantel-Haenszel = prior anti-TNF versus anti-TNF-naive

7. Secondary Outcome: Proportion of Participants Who Achieved Mucosal Healing at Week 8
Description: Mucosal healing is defined as an Endoscopy Subscore of 0 or 1 as assessed by flexible sigmoidoscopy. Possible scores range from 0-3 as follows:
  0 = Normal or inactive disease, 1 = Mild disease (erythema, decreased vascular pattern, mild friability), 2 = Moderate disease (marked erythema, absent vascular pattern, friability, erosions), 3 = Severe disease(spontaneous bleeding, ulceration).
Time Frame: Week 8
Population: as for outcome 3
Measure: Number; unit: Percentage of Participants
Arm/Group | Adalimumab 160/80/40 | Placebo
Number analyzed (Participants) | 248 | 246
Percentage of Participants | 41.1 | 31.7
Statistical Analysis 1: Comparison: Adalimumab 160/80/40 vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.032, Cochran-Mantel-Haenszel — Testing of ranked secondary measures was only started if significant group differences existed for both co-primary measures. Significant results for higher-ranked measure were needed to test next lower-ranked measure to control for multiple testing; Stratification levels for Cochran-Mantel-Haenszel = prior anti-TNF versus anti-TNF-naive

8. Secondary Outcome: Proportion of Participants Who Achieved Mucosal Healing at Week 52
Description: as for outcome 7
Time Frame: Week 52
Population: as for outcome 3
Measure: Number; unit: Percentage of Participants
Arm/Group | Adalimumab 160/80/40 | Placebo
Number analyzed (Participants) | 248 | 246
Percentage of Participants | 25.0 | 15.4
Statistical Analysis 1: Comparison: Adalimumab 160/80/40 vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.009, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; Stratification levels for Cochran-Mantel-Haenszel = prior anti-TNF versus anti-TNF-naive

9. Secondary Outcome: Proportion of Participants Who Achieved Sustained Mucosal Healing at Both Week 8 and Week 52
Description: as for outcome 7
Time Frame: Week 8, Week 52
Population: as for outcome 3
Measure: Number; unit: Percentage of Participants
Arm/Group | Adalimumab 160/80/40 | Placebo
Number analyzed (Participants) | 248 | 246
Percentage of Participants | 18.5 | 10.6
Statistical Analysis 1: Comparison: Adalimumab 160/80/40 vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.013, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; Stratification levels for Cochran-Mantel-Haenszel = prior anti-TNF versus anti-TNF-naive

10. Secondary Outcome: Proportion of Participants Who Discontinued Corticosteroid Use Before Week 52 and Achieved Clinical Remission Per Mayo Score at Week 52
Description: as for outcome 2
Time Frame: Baseline to Week 52
Population: as for outcome 3
Measure: Number; unit: Percentage of Participants
Arm/Group | Adalimumab 160/80/40 | Placebo
Number analyzed (Participants) | 150 | 140
Percentage of Participants | 13.3 | 5.7
Statistical Analysis 1: Comparison: Adalimumab 160/80/40 vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.035, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; Stratification levels for Cochran-Mantel-Haenszel = prior anti-TNF versus anti-TNF-naive

11. Secondary Outcome: Proportion of Participants With Physician's Global Assessment Subscore Indicative of Mild Disease (a Score of 0 or 1) at Week 8
Description: The PGA includes the 3 other subscores (SFS, RBS, and Endoscopy), the participant's daily record of abdominal discomfort and functional assessment, and other observations such as physical findings and the participant's performance status. Possible scores range from 0-3 as follows:
  0 = Normal (other subscores are 0), 1 = Mild disease (other subscores are mostly 1), 2 = Moderate disease (other subscores are 1 to 2), 3 = Severe disease (other subscores are 2 to 3).
Time Frame: Week 8
Population: as for outcome 3
Measure: Number; unit: Percentage of Participants
Arm/Group | Adalimumab 160/80/40 | Placebo
Number analyzed (Participants) | 248 | 246
Percentage of Participants | 46.0 | 37.4
Statistical Analysis 1: Comparison: Adalimumab 160/80/40 vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.058, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; Stratification levels for Cochran-Mantel-Haenszel = prior anti-TNF versus anti-TNF-naive

12. Secondary Outcome: Proportion of Participants With Stool Frequency Subscore Indicative of Mild Disease (a Score of 0 or 1) at Week 8
Description: SFS ranges from 0-3 as follows:
  0 = Normal number of stools for this participant, 1 = 1-2 stools more than normal, 2 = 3-4 stools more than normal, 3 = 5 or more stools more than normal. The participant served as his/her own control.
Time Frame: Week 8
Population: as for outcome 3
Measure: Number; unit: Percentage of Participants
Arm/Group | Adalimumab 160/80/40 | Placebo
Number analyzed (Participants) | 248 | 246
Percentage of Participants | 37.9 | 28.5
Statistical Analysis 1: Comparison: Adalimumab 160/80/40 vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.028, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; Stratification levels for Cochran-Mantel-Haenszel = prior anti-TNF versus anti-TNF-naive

13. Secondary Outcome: Proportion of Participants With Rectal Bleeding Subscore Indicative of Mild Disease (a Score of 0 or 1) at Week 8
Description: RBS ranges from 0-3 as follows:
  0 = no blood seen, 1 = streaks of blood with stool less than half the time, 2 = obvious blood with stool most of the time, 3 = blood alone passed
Time Frame: Week 8
Population: as for outcome 3
Measure: Number; unit: Percentage of Participants
Arm/Group | Adalimumab 160/80/40 | Placebo
Number analyzed (Participants) | 248 | 246
Percentage of Participants | 70.2 | 58.1
Statistical Analysis 1: Comparison: Adalimumab 160/80/40 vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.006, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; Stratification levels for Cochran-Mantel-Haenszel = prior anti-TNF versus anti-TNF-naive

14. Secondary Outcome: Proportion of Participants Who Discontinued Corticosteroid Use for At Least 90 Days and Achieved Clinical Remission Per Mayo Score at Week 52
Description: as for outcome 2
Time Frame: Baseline to Week 52
Population: as for outcome 3
Measure: Number; unit: Percentage of Participants
Arm/Group | Adalimumab 160/80/40 | Placebo
Number analyzed (Participants) | 150 | 140
Percentage of Participants | 13.3 | 5.7
Statistical Analysis 1: Comparison: Adalimumab 160/80/40 vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.035, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; Stratification levels for Cochran-Mantel-Haenszel = prior anti-TNF versus anti-TNF-naive

15. Secondary Outcome: Proportion of Participants Who Discontinued Corticosteroid Use and Achieved Clinical Remission Per Mayo Score (Sustained) at Both Weeks 32 and 52
Description: as for outcome 2
Time Frame: Week 32, Week 52
Population: as for outcome 3
Measure: Number; unit: Percentage of Participants
Arm/Group | Adalimumab 160/80/40 | Placebo
Number analyzed (Participants) | 150 | 140
Percentage of Participants | 10.0 | 1.4
Statistical Analysis 1: Comparison: Adalimumab 160/80/40 vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.002, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; Stratification levels for Cochran-Mantel-Haenszel = prior anti-TNF versus anti-TNF-naive

16. Secondary Outcome: Proportion of Inflammatory Bowel Disease Questionnaire Responders at Week 52
Description: Response per the Inflammatory Bowel Disease Questionnaire (IBDQ) was defined as at least a 16-point increase from Baseline in total IBDQ score. The IBDQ is a 32-item questionnaire consisting of 4 dimensions: bowel-related symptoms, systemic function, social function, and emotional status. The responses to questions within each domain range from 1 (significant impairment) to 7 (no impairment), with total score ranging from 32 (very poor) to 224 (perfect health-related quality of life).
Time Frame: Week 52
Population: as for outcome 3
Measure: Number; unit: Percentage of Participants
Arm/Group | Adalimumab 160/80/40 | Placebo
Number analyzed (Participants) | 248 | 246
Percentage of Participants | 26.2 | 16.3
Statistical Analysis 1: Comparison: Adalimumab 160/80/40 vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.007, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; Stratification levels for Cochran-Mantel-Haenszel = prior anti-TNF versus anti-TNF-naive

17. Secondary Outcome: Proportion of Inflammatory Bowel Disease Questionnaire Responders at Week 8
Description: as for outcome 16
Time Frame: Week 8
Population: as for outcome 3
Measure: Number; unit: Percentage of Participants
Arm/Group | Adalimumab 160/80/40 | Placebo
Number analyzed (Participants) | 248 | 246
Percentage of Participants | 58.1 | 45.5
Statistical Analysis 1: Comparison: Adalimumab 160/80/40 vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.006, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; Stratification levels for Cochran-Mantel-Haenszel = prior anti-TNF versus anti-TNF-naive

ADVERSE EVENTS:
Time Frame: Double-Blind (DB) period: From 1st study drug dose in DB period to 70 days after last DB study drug dose or until switch to Open-Label. Any Adalimumab: From 1st adalimumab dose up 70 days after last adalimumab dose or until switch to extension study.
Description: **518 participants were randomized into the study; 1 subject did not receive study drug and was excluded from the safety analyses. The number of participants in the Safety population (at least 1 dose of study drug) was higher (517) than that in the ITT population (494), as the latter excluded participants from 3 non-compliant clinical sites.**
Groups:
- Adalimumab Group - Double-Blind Period: During the Double-Blind period, the Adalimumab treatment group received a dose of 160 mg at Week 0, 80 mg at Week 2, and 40 mg every other week (eow) starting at Week 4 (160/80/40 mg).
- Placebo Group - Double-Blind Period: The placebo treatment group received placebo throughout the Double-Blind period.
- Any Adalimumab: During the Double-Blind period, only the Adalimumab treatment group received active study drug (dose of 160 mg at Week 0, 80 mg at Week 2, and 40 mg every other week (eow) starting at Week 4 [160/80/40 mg]). After the switch to open-label treatment, participants in both treatment groups received adalimumab 40 mg eow, unless they dose-escalated, in which case they received adalimumab 40 mg every week (ew). Consequently, this analysis set combined adalimumab exposure from both the Double-Blind and Open-Label periods.
Arm/Group | Adalimumab Group - Double-Blind Period | Placebo Group - Double-Blind Period | Any Adalimumab
Serious Adverse Events (participants affected / at risk) | 31/257 | 32/260 | 61/398
Other Adverse Events (participants affected / at risk) | 139/257 | 142/260 | 204/398
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab Group - Double-Blind Period (N=257) | Placebo Group - Double-Blind Period (N=260) | Any Adalimumab (N=398)
Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 3
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 2
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 1
Anal fistula (Gastrointestinal disorders) | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 16 | 18 | 35
Constipation (Gastrointestinal disorders) | 1 | 0 | 1
Gastrointestinal dysplasia (Gastrointestinal disorders) | 1 | 0 | 1
Crohn's disease (Gastrointestinal disorders) | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 2
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 0 | 1
Localized intraabdominal fluid collection (Gastrointestinal disorders) | 1 | 0 | 1
Obstruction gastric (Gastrointestinal disorders) | 1 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Rectal perforation (Gastrointestinal disorders) | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 1
Anal abscess (Infections and infestations) | 1 | 1 | 1
Appendicitis (Infections and infestations) | 1 | 0 | 2
Catheter sepsis (Infections and infestations) | 1 | 0 | 1
Cytomegalovirus colitis (Infections and infestations) | 0 | 1 | 1
Erysipelas (Infections and infestations) | 0 | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 0 | 1
Liver abscess (Infections and infestations) | 0 | 1 | 0
Perineal abscess (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Pneumonia necrotizing (Infections and infestations) | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Salmonellosis (Infections and infestations) | 1 | 0 | 1
Scrotal abscess (Infections and infestations) | 0 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 1 | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Ligament calcification (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Abortion (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 1 | 1 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1
Cystocele (Reproductive system and breast disorders) | 0 | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1
Organizing pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 1 | 1
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 0 | 4 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 1 | 2
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 0
Thrombophlebitis superficial (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab Group - Double-Blind Period (N=257) | Placebo Group - Double-Blind Period (N=260) | Any Adalimumab (N=398)
Anaemia (Blood and lymphatic system disorders) | 8 | 14 | 21
Abdominal pain (Gastrointestinal disorders) | 19 | 16 | 27
Colitis ulcerative (Gastrointestinal disorders) | 42 | 58 | 71
Nausea (Gastrointestinal disorders) | 15 | 22 | 23
Fatigue (General disorders) | 16 | 15 | 25
Pyrexia (General disorders) | 11 | 14 | 23
Nasopharyngitis (Infections and infestations) | 45 | 27 | 68
Upper respiratory tract infection (Infections and infestations) | 11 | 14 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 20 | 16 | 30
Headache (Nervous system disorders) | 22 | 37 | 31
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 15 | 7 | 23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.